CLINICAL TRIAL: NCT03936335
Title: Dupilumab and Pregnancy Outcomes: A Retrospective Cohort Study Using Administrative Healthcare Databases (Dupi PODS)
Brief Title: An Observational Retrospective Cohort Study Being Conducted in Women With Atopic Dermatitis (AD)
Status: Recruiting | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: R668-AD-1760; 43838 (Registry Identifier: EU HMA-EMA Catalogue)
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Adverse Pregnancy Outcomes; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dupilumab cohort: Exposed to dupilumab during the relevant exposure window:
  * First trimester
  * Pregnancy
  Interventions: Drug: dupilumab
- Other systemic therapy or phototherapy cohort: Exposed to systemic medications other than dupilumab or to phototherapy during the relevant exposure window:
  * First trimester
  * Pregnancy
- Unexposed cohort: * Not exposed to systemic medications (including dupilumab) or phototherapy; and
  * Received topical prescription therapy, or a second diagnosis for AD on a date that differs from the base population qualifying AD diagnosis date during the relevant exposure window:
  * First trimester
  * Pregnancy

INTERVENTIONS:
Drug: dupilumab — No study drug will be administered. This study is based on an analysis of automated medical and prescription claims, supplemented by information abstracted from the medical record.
  Other Names: REGN668; Dupixent®; SAR23189
  Groups: Dupilumab cohort

SUMMARY:
The objective of this study is to describe and compare the incidence of adverse pregnancy outcomes (spontaneous abortion/miscarriage, stillbirth) and prevalence of adverse infant outcomes (major congenital malformations [MCMs], small for gestational age [SGA]) in women with AD who are treated with dupilumab during pregnancy relative to women with AD who are not treated with dupilumab during pregnancy.

ELIGIBILITY:
Key Inclusion Criteria:

* Continuous medical and pharmacy benefit coverage for at minimum 6 months prior to and including the estimated LMP
* Diagnosis code indicative of AD in the period from up to 1 year prior to the estimated LMP through the end of the pregnancy

Note: Other Protocol Defined Inclusion / Exclusion Criteria Apply

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Adult women with AD who are pregnant between 01 April 2017 and 31 March 2024 (with the start of pregnancy to be defined by the estimated last menstrual period (LMP))
Sampling Method: Non-Probability Sample
Enrollment: 3930 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2027-01-21 (Estimated); Study Completion 2027-01-21 (Estimated)

PRIMARY OUTCOMES:
Prevalence of MCMs | Up to 21 months
  Initially identified through the presence of corresponding codes on the insurance claims, confirmed through medical record review for infant outcomes: 01 April 2017 through December 2024

SECONDARY OUTCOMES:
Incidence of spontaneous abortion or miscarriage | Up to 9 months
  Identified through the presence of corresponding codes on the insurance claims for pregnancy outcomes: 01April 2017 through 31 March 2024
Incidence of stillbirth | Up to 9 months
  Identified through the presence of corresponding codes on the insurance claims for pregnancy outcomes: 01April 2017 through 31 March 2024
Incidence of SGA | Up to 21 months
  Identified through the presence of corresponding codes on the insurance claims for infant outcomes: 01 April 2017 through December 2024

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Research Site, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No